CLINICAL TRIAL: NCT01056289
Title: A Randomized, Double-Blind, Parallel Group Study To Compare Discontinuation Symptoms In Abrupt Discontinuation Versus A 1-Week Tapering Regimen In Subjects With MDD Treated For 24 Weeks With Open-Label 50 mg DVS SR Formulation
Brief Title: Study Comparing Discontinuation Symptoms Of DVS SR In Subjects With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-4437; B2061010
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2011-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desvenlafaxine Succinate Sustained-Release Formulation 50 mg (Active Comparator)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release Formulation 50 mg
- Desvenlafaxine Succinate Sustained-Release Formulation 25 mg (Active Comparator)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release Formulation 25 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release Formulation 50 mg — DVS SR 50 mg Reference Group/Arm, oral tablet, 2 tablets/day during the first week and 1 tablet/day during weeks 2 through 4 of the double-blind treatment phase.
  Arms: Desvenlafaxine Succinate Sustained-Release Formulation 50 mg
Drug: Desvenlafaxine Succinate Sustained-Release Formulation 25 mg — DVS SR 25 mg Taper Group/Arm, oral tablet, 2 tablets/day during the first week and 1 tablet/day during weeks 2 through 4 of the double-blind treatment phase.
  Arms: Desvenlafaxine Succinate Sustained-Release Formulation 25 mg
Drug: Placebo — DVS SR Placebo Abrupt Discontinuation Group/Arm, oral tablet, 2 tablets/day during the first week and 1 tablet/day during weeks 2 through 4 of the double-blind treatment phase.
  Arms: Placebo

SUMMARY:
Study Comparing Discontinuation Symptoms in subjects with Major Depressive Disorder treated for 24 Weeks with Open-label 50 mg Desvenlafaxine Succinate Sustained-Release Formulation (DVS SR)

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of Major Depressive Disorder
* Hamilton Psychiatric Rating Scale for Depression-17-Item score of greater than or equal to 14 at baseline

Exclusion Criteria:

* Current psychoactive substance abuse or dependence, manic episode, or a lifetime diagnosis of bipolar or psychotic disorder
* Potentially violent to others or is at significant risk for suicide
* History or current evidence of gastrointestinal disease or history of surgery known to interfere with absorption or excretion
* Known presence of raised intraocular pressure or history of narrow angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Ninan PT, Musgnung J, Messig M, Buckley G, Guico-Pabia CJ, Ramey TS. Incidence and Timing of Taper/Posttherapy-Emergent Adverse Events Following Discontinuation of Desvenlafaxine 50 mg/d in Patients With Major Depressive Disorder. Prim Care Companion CNS Disord. 2015 Feb 5;17(1):10.4088/PCC.14m01715. doi: 10.4088/PCC.14m01715. eCollection 2015. PMID 26137358
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-4437&StudyName=Study%20Comparing%20Discontinuation%20Symptoms%20Of%20DVS%20SR%20In%20Subjects%20With%20Major%20Depressive%20Disorder%20%28MDD%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants entered a 24 Week Open-label treatment phase; participants who completed the Open-label phase were randomized to a 4 Week Double-blind treatment phase.
Groups:
- DVS SR 50 mg (Open-label Phase): Desvenlafaxine Succinate Sustained-Release Formulation (DVS SR) 50 milligrams (mg) by mouth (PO) once daily (QD) for 24 Weeks.
- DVS SR 50 mg (Double-blind Phase): DVS SR 50 mg (reference group): 2 tablets PO once daily (QD) for 1 week (1 tablet DVS SR 50 mg and 1 tablet placebo 25 mg) then DVS SR 50 mg 1 tablet PO QD Weeks 2 through 4.
- DVS SR 25 mg (Double-blind Phase): DVS SR 25 mg (taper group): 2 tablets PO QD for 1 week (1 tablet placebo 50 mg and 1 tablet DVS SR 25 mg) then placebo 50 mg 1 tablet PO QD Weeks 2 through 4.
- Placebo (Double-blind Phase): Placebo (abrupt-discontinuation group): 2 tablets PO QD for 1 week (1 tablet placebo 50 mg and 1 tablet placebo 25 mg) then placebo 50 mg 1 tablet PO QD Weeks 2 through 4.
Period: Open-label Phase
Arm/Group | DVS SR 50 mg (Open-label Phase) | DVS SR 50 mg (Double-blind Phase) | DVS SR 25 mg (Double-blind Phase) | Placebo (Double-blind Phase)
Started | 480 | 0 | 0 | 0
Completed | 361 (Participants transitioned to Double-blind phase) | 0 | 0 | 0
Not Completed | 119 | 0 | 0 | 0
Not completed — Adverse Event | 29 | 0 | 0 | 0
Not completed — Lost to Follow-up | 30 | 0 | 0 | 0
Not completed — Other | 9 | 0 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 0 | 0 | 0
Not completed — Lack of Efficacy | 18 | 0 | 0 | 0
Not completed — Not randomized to Double-blind phase | 1 | 0 | 0 | 0
Period: Double-blind Phase
Arm/Group | DVS SR 50 mg (Open-label Phase) | DVS SR 50 mg (Double-blind Phase) | DVS SR 25 mg (Double-blind Phase) | Placebo (Double-blind Phase)
Started | 0 | 73 | 140 | 148
Completed | 0 | 69 | 127 | 138
Not Completed | 0 | 4 | 13 | 10
Not completed — Adverse Event | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 2 | 2
Not completed — Other | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 2
Not completed — Discontinuation symptom | 0 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: 24 Week Open-label phase DVS SR 50 mg PO QD followed by 4 Week Double-blind phase: DVS SR 50 mg (reference group), DVS SR 25 mg (taper group), or Placebo (abrupt-discontinuation group).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 480
Age Continuous [Mean (Standard Deviation); unit: years] | 46.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330
  Male | 150

OUTCOME MEASURES:

1. Primary Outcome: Total Discontinuation - Emergent Signs and Symptoms (DESS) Score Over the First 2 Weeks of the Double-blind Phase
Description: Clinician-administered 43-item assessment to evaluate discontinuation-emergent symptoms resulting from withdrawal from study treatment. Total score=sum of number of new symptoms and old (but worse) symptoms (score=1) and old and unchanged symptom, absent, or old symptom but improved (score=0); total possible range 0 to 43. Higher score=more symptoms. New symptom=any symptom that appeared within 7 days before DESS administration; old symptom=any symptom that appeared 7 days before DESS administration and continued into 7-day period. DESS calculated as 2*mean(of DESSDB Week 1, DESSDB Week 2).
Time Frame: Double-blind phase: Week 1 (Study Day 175), Week 2 (Study Day 182)
Population: Full Analysis Set (FAS): all randomized participants who had at least 1 postrandomization DESS record. Mean was adjusted for baseline DESS score and study center.
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- DVS SR 50 mg: DVS SR 50 mg (reference group): 2 tablets PO once daily (QD) for 1 week (1 tablet DVS SR 50 mg and 1 tablet placebo 25 mg) then DVS SR 50 mg 1 tablet PO QD Weeks 2 through 4.
- DVS SR 25 mg: DVS SR 25 mg (taper group): 2 tablets PO QD for 1 week (1 tablet placebo 50 mg and 1 tablet DVS SR 25 mg) then placebo 50 mg 1 tablet PO QD Weeks 2 through 4.
- Placebo: Placebo (abrupt-discontinuation group): 2 tablets PO QD for 1 week (1 tablet placebo 50 mg and 1 tablet placebo 25 mg) then placebo 50 mg 1 tablet PO QD Weeks 2 through 4.
Arm/Group | DVS SR 50 mg | DVS SR 25 mg | Placebo
Number analyzed (Participants) | 72 | 139 | 146
scores on a scale | 4.1 (0.72) | 4.8 (0.54) | 5.3 (0.52)
Statistical Analysis 1: Comparison: DVS SR 50 mg vs Placebo; Difference: Placebo versus DVS SR 50 mg; Test type: Non-Inferiority or Equivalence — Null hypothesis: absolute difference between the 2 discontinuation regimens in DESS total scores was >2.5. Alternative hypothesis: absolute difference was ≤2.5; tested by calculating 95% 2-sided confidence intervals (CIs) on the mean difference between the 2 regimens. If absolute values of both confidence limits were ≤2.5, then the regimens were declared equivalent; ANCOVA; Mean Difference (Final Values) = 1.16, 95% CI 2-sided [-0.51 to 2.83]
Statistical Analysis 2: Comparison: DVS SR 50 mg vs DVS SR 25 mg; Difference: DVS SR 25 mg versus DVS SR 50 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-1.03 to 2.35]
Statistical Analysis 3: Comparison: DVS SR 25 mg vs Placebo; Difference: Placebo versus DVS SR 25 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.88 to 1.89]

2. Secondary Outcome: Percentage of Participants With Taper Adverse Events (AEs) in the Double-blind Phase
Description: Any untoward medical occurrence in a patient who received study drug was considered an AE without regard to possibility of causal relationship. Taper-emergent AEs (TPAEs) are those events which occurred during the double-blind period but did not occur during the last 7 days of the on-therapy period or existed during the last 7 days and worsened in the double-blind period.
Time Frame: Double-blind phase: Baseline (Study Day 168) up to Week 4 (Study Day 196)
Population: Safety population (Double-blind phase): all participants who received at least 1 dose of study treatment and were randomized into the Double-blind treatment phase.
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR 50 mg | DVS SR 25 mg | Placebo
Number analyzed (Participants) | 73 | 140 | 148
percentage of participants | 35.6 | 38.6 | 50.7

3. Secondary Outcome: Percentage of Participants Who Were Unable to Successfully Complete Tapering of the Study Drug Because of the Number and/or Severity of Their Discontinuation Symptoms
Description: Discontinuation symptoms may occur following abrupt cessation of serotonergic antidepressants in a minority of participants following short-term treatment of an episode of Major Depressive Disorder (MDD). The symptoms include emotional and somatic symptoms such as dizziness, nausea, and paresthesia and typically appear within 2 to 3 days of reducing the dose or stopping the antidepressant medication. Discontinuation symptoms are usually mild and resolve spontaneously within a week in the majority of patients, though a minority can have intense and prolonged symptoms.
Time Frame: Double-blind phase: Baseline (Study Day 168) up to Week 4 (Study Day 196)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR 50 mg | DVS SR 25 mg (Double-blind Phase) | Placebo
Number analyzed (Participants) | 72 | 139 | 146
percentage of participants | 1.4 | 1.4 | 1.4

ADVERSE EVENTS:
Time Frame: Events collected from the signing of the informed consent form up to 14 days after the last dose of study treatment
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- DVS SR 50 mg (Open-label Phase): DVS SR 50 mg PO QD for 24 Weeks.
Arm/Group | DVS SR 50 mg (Open-label Phase) | DVS SR 50 mg (Double-blind Phase) | DVS SR 25 mg (Double-blind Phase) | Placebo (Double-blind Phase)
Serious Adverse Events (participants affected / at risk) | 5/480 | 0/73 | 0/140 | 0/148
Other Adverse Events (participants affected / at risk) | 197/480 | 9/73 | 18/140 | 33/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 mg (Open-label Phase) (N=480) | DVS SR 50 mg (Double-blind Phase) (N=73) | DVS SR 25 mg (Double-blind Phase) (N=140) | Placebo (Double-blind Phase) (N=148)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 mg (Open-label Phase) (N=480) | DVS SR 50 mg (Double-blind Phase) (N=73) | DVS SR 25 mg (Double-blind Phase) (N=140) | Placebo (Double-blind Phase) (N=148)
Diarrhoea (Gastrointestinal disorders) | 25 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 28 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 64 | 5 | 6 | 9
Fatigue (General disorders) | 24 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 25 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 39 | 1 | 8 | 14
Headache (Nervous system disorders) | 52 | 3 | 10 | 20
Insomnia (Psychiatric disorders) | 38 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.